CLINICAL TRIAL: NCT06283329
Title: Residual Vocal Cords Curarization Correlation Between Clinical and Ultrasound Endpoints
Status: Completed | Type: Observational
Sponsor: General Administration of Military Health, Tunisia (Network)
Responsible Party: Principal Investigator, Hedi Gharsallah, Professor, General Administration of Military Health, Tunisia
Other Study IDs: echographic VC curarization
Record Dates: First submitted 2024-02-15; First posted 2024-02-28 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Residual Curarization
Keywords: residual curarization; airway access; echography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group A: a group of patients receiving systematic decurarization using neostigmine , a unique dose of 40 µg/kg associated with atropine 20 µg/kg
  Interventions: Diagnostic Test: vocal cords echography
- Group B: a group of patients extubated through clinical criteria without use of neostigmine
  Interventions: Diagnostic Test: vocal cords echography

INTERVENTIONS:
Diagnostic Test: vocal cords echography — Ultrasound assessments of the amplitude of the vocal cords movement were performed on a sagittal median section of the arytenoid cartilages with a 30° inclination using a Golf Head ultrasound probe at 3 different time points: before induction (T0), after extubation (T1), in recovery room 30 minutes after extubation(T2). We have defined H0, H1 and H2, the maximum course of the vocal cords measured respectively at T0, T1 and T2

SUMMARY:
Through recent studies residual curarization (RC) remains frequent but serious event, that could be easily avoided in the presence of a paraclinical monitoring and by antagonization of curares. However, conventional monitors focus only on peripheral muscles, whereas ultrasonography allows direct visualization of laryngeal muscles, particularly the vocal cords, which are directly influenced by neuromuscular blocking agents. The aim of the study was to evaluate the ultrasound mobility of the vocal cords after awakening and extubation of general anesthesia compared to their preoperative mobility and its correlation with clinical and paraclinical diagnostic criteria (DG) for RC.

DETAILED DESCRIPTION:
The investigators conducted an analytical prospective observational and comparative study between March 2022 and May 2022. The investigators included all patients proposed for elective surgery under general anesthesia with Tracheal intubation other than ENT surgery, ages 18 to 70 years, consenting, classified ASA class I, II, or III, with no history of difficult intubation and/or ventilation, divided into two groups that differ by neostigmine use: group A: systematic decurarization, group B: extubation through clinical criteria. Ultrasound assessments of the vocal cords were performed at 3 different time points: before induction (T0), after extubation (T1), in SSPI 30 minutes after extubation (T2). The investigators have defined H0, H1 and H2, the maximum amplitudes of the vocal cords measured respectively at T0, T1 and T2. The primary endpoint was the ultrasound judged vocal cord range of motion with a ratio of pre- to post curarization amplitude defining the HA score, calculated using the following formulas: H0-H1, H0-H2, HAt1=H1/H0, HAt2=H2/H0. The investigators conducted a single then multi-variate analysis.

ELIGIBILITY:
Inclusion Criteria:

* patients proposed for elective surgery under general anesthesia with Tracheal intubation other than ENT surgery

Exclusion Criteria:

* Patients whose airway management was ensured by supraglottic device
* Patients who have experienced an intraoperative incident requiring them to be kept intubated after surgery
* ENT surgery
* non consenting patients

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: patients proposed for elective surgery under general anesthesia with Tracheal intubation other than ENT surgery, ages 18 to 70 years, consenting, classified ASA class I, II, or III with no history of difficult intubation and/or ventilation,
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2023-12-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Echographic mobility of vocal cords at different times in post extubation | before induction (T0), immediately after extubation (T1) and 30 minutes after extubation (T2)
  measured in TM mode, mobility will be measured in millimeters from baseline curve

CONTACTS AND LOCATIONS:
Locations (1):
- Elaskri Haythem, Tunis, Tunisia

IPD SHARING:
Plan to Share IPD: Undecided